CLINICAL TRIAL: NCT02786407
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Botulinum Toxin Type A for Injection in Chinese Subjects With Overactive Bladder (OAB)
Brief Title: A Study to Evaluate the Efficacy and Safety of Botulinum Toxin Type A in Patients With Overactive Bladder (OAB)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HengLi004
Record Dates: First submitted 2016-05-17; First posted 2016-06-01 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; Botulinum Toxin Type A for Injection
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Injections; Hengli BTX-A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum Toxin Type A for Injection (Active Comparator): Botulinum Toxin Type A is a specific formulation of a locally injected muscle relaxant whose active ingredient is botulinum toxin type A produced by clostridium botulinum A strain Hall. Excipients contain sucrose,dextran and gelatin.
  Interventions: Drug: Botulinum Toxin Type A for Injection
- Placebo (Placebo Comparator): The placebo does not include botulinum toxin A ,but include sucrose,dextran and gelatin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A for Injection — In these studies,patients received a minimum intramuscular(IM) dose of 100U of Botulinum Toxin Type A administered to 20 injection sites
  Other Names: HengLi®
  Arms: Botulinum Toxin Type A for Injection
Drug: Placebo — In these studies,patients received placebo administered to 20 injection sites
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study designed to evaluate the efficacy and safety of Botulinus Toxin Type A for Injection (HengLi®) in patients with overactive bladder (OAB) . Approximately 216 subjects will be enrolled. Subjects will be randomized 2:1 to receive intradetrusor injection of Botulinus Toxin Type A for Injection (HengLi®) 100 U or placebo. The study contains two parts: core double-blinded phase and extension phase. In the core double-blinded phase, eligible subjects must attend three study visits posttreatment 12 weeks. During the extension phase, subjects must also attend three study visits (12 weeks). The primary efficacy variables is the change from baseline in the daily average frequency of micturition at week 6 after the first treatment.A 3-day paper bladder diary will be used before each study visits (screening period, the second week, the sixth week, the twelfth week, the fourteenth week, the eighteenth week and the twenty fourth week ) to collect all OAB symptoms (episodes of urgency, incontinence, micturition and nocturia) and volume per voidSafety parameters will also be measured, including adverse events, vital signs (pulse and blood pressure) and clinical laboratory tests (haematology, serum chemistry and urinanalysis).

DETAILED DESCRIPTION:
Eligible patients will be randomized on day 1 to receive double-blind treatment with Botulinus Toxin Type A for Injection (HengLi®) 100U or placebo in a 2:1 ratio. A total of 216 subjects will be randomized into this study. Followup visits will occur at day 0, week 6 and 12, and week 14, 18 and 24 thereafter until study exit at week 24 unless re-treatment was necessary. The primary efficacy variables is the change from baseline in the daily average frequency of micturition at week 6. After a screening period of 1 week, all eligible patients will be randomized to receive a single intramuscular treatment with Botulinus Toxin Type A for Injection (HengLi®) or placebo at day 0 (visit 0).

ELIGIBILITY:
Inclusion Criteria:

1. All patients should provided written informed consent.
2. Patients with idiopathic or neurogenic overactive bladder with symptoms of episodes of urgency, incontinence, micturition and nocturia,( maintaining spontaneous voiding ).
3. Patients must experienced 3 or more urgency UI episodes in a 3-day period and an average of 8 or moremicturitions per day.
4. Patients were inadequately treated with prior anticholinergic therapy due to inadequate efficacy or intolerable side effects.
5. Anticholinergic use was not permitted within 7 days of screening or patients treated with anticholinergics at baseline continued at a stable dose throughout the study.

Exclusion Criteria:

1. Patients with difficulty urinating have a PVR of 50 ml or more.
2. Patients requiring indwelling catheter or clean intermittent catheterization (CIC).
3. Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
4. People who are allergic to study drugs or its ingredients or allergic should be excluded.
5. Current severe cardiovascular disease ongoing clinical instability.
6. Renal insufficiency and serum creatinine greater than 1.5 times the upper limit of normal.
7. Liver diseases, ALT or AST greater than 2 times the upper limit of normal.
8. Alcohol or drug abusers.
9. Have participated in the clinical trials of other drugs within a month.
10. Any previous botulinum toxin therapy for a urologic condition within 6 months.
11. Urinary tract infection (① patients with symptoms of fever, pyuria, urinary frequency, urgency or dysuria etc.; ② positive urine culture ( bacterial colony counts > 10^5 cfu/ml) or urine WBC> 10/ HPF; meet both of ① and ② or any one can be diagnosed as a urinary tract infection).
12. Patients accompany of bladder stones, ureteral stones or urethral; or lithotripsy performed within 3 months.
13. Patients of bladder or prostate cancer.
14. Patients with diabetes.
15. Patients with aminoglycoside antibiotics or neuromuscular junction function drugs within one week.
16. Any medical condition that may lead the subject to increased risk with exposure to Botulinum Toxin Type A, including myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other disorder that might have interfered with neuromuscular function.
17. Patients with bleeding tendency.
18. Patients have used anticoagulant agents within one week before the first use of study drug.
19. Investigator's opinion that the subject has a concurrent condition(s) that may put the subject at significant risk, may confound the study results, or may interfere significantly with the conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
average frequency of micturition | Baseline(week -1 to 0)and core phase(week 6)
  The primary efficacy variables is the change from baseline in the daily average frequency of micturition at week 6 after the first treatment.

SECONDARY OUTCOMES:
The change from baseline in the daily average frequency of urgency episodes and the scores. | Baseline and Week 2,6,12,14,18,24
  The degree of urgency is divided into 5 grades (With 0 points representing no hurry, hurry on behalf of 5 points, 1~5 points gradually increase depending on the degree of urgency)
average frequency of UI episodes | Baseline and Week 2,6,12,14,18,24
  The change from baseline in the daily average frequency of UI episodes
volume per micturition | Baseline and Week 2,6,12,14,18,24
  The change from baseline in volume voided per micturition
maximum cystometric capacity (MCC) | Baseline(week -1 to 0)and core phase(week 6)
  The change from baseline in MCC at week 6 after the first treatment ( Only in patients with neurogenic overactive bladder )
maximum detrusor pressure during first involuntary detrusor contraction (PdetmaxIDC) | Baseline(week -1 to 0)and core phase(week 6)
  The change from baseline in PdetmaxIDC at week 6 after the first treatment ( Only in patients with neurogenic overactive bladder )
volume at first IDC (VPmaxIDC) | Baseline(week -1 to 0)and core phase(week 6)
  The change from baseline in VPmaxIDC at week 6 after the first treatment ( Only in patients with neurogenic overactive bladder )
The change from baseline in the QOL score | Baseline and Week 2,6,12,14,18,24
  The change from baseline in the QOL score
The change from baseline in the OABSS total summary score | Baseline and Week 2,6,12,14,18,24
  The change from baseline in the OABSS total summary score

IPD SHARING:
Plan to Share IPD: No